CLINICAL TRIAL: NCT00943956
Title: A Phase I Trial to Evaluate Acute and Late Toxicities of Concurrent Treatment With Everolimus (RAD001) and Radio-Hormonotherapy in High-risk Prostate Cancer.(RHOMUS)
Brief Title: Everolimus, Bicalutamide, and Leuprolide Acetate in Treating Patients Undergoing Radiation Therapy For High-Risk Locally Advanced Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000639358; CLCC-RHOMUS; CRAD001 C2486; INCA-RECF0921; EUDRACT-2007-003620-38
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Prostate Cancer
Keywords: stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Everolimus; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus (Experimental): Everolimus + radiation
  Interventions: Drug: bicalutamide; Drug: everolimus; Drug: leuprolide acetate; Radiation: external beam radiation therapy

INTERVENTIONS:
Drug: bicalutamide
Drug: everolimus
Drug: leuprolide acetate
Radiation: external beam radiation therapy

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as bicalutamide and leuprolide acetate may lessen the amount of androgens made by the body. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving everolimus together with bicalutamide, leuprolide acetate, and radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of everolimus when given together with bicalutamide and leuprolide acetate in treating patients with high-risk locally advanced prostate cancer undergoing radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess acute and late toxicities in patients with high-risk, locally advanced prostate cancer.

Secondary

* To assess the biochemical-free survival of these patients.
* To assess metastasis-free survival of these patients.
* To assess the overall survival of these patients.
* To assess the molecular characteristics of the tumor before treatment and correlate with outcomes.

OUTLINE: This is a dose-escalation study of everolimus.

Patients undergo radiotherapy to the prostate and seminal vesicles once daily, 5 days a week, for 7.5 weeks.

Beginning the week before radiotherapy, patients receive oral bicalutamide once daily for 1 month and oral everolimus twice daily for 8.5 weeks. Beginning on the first week of radiotherapy, patients receive leuprolide acetate subcutaneously every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of high-risk, locally advanced prostate cancer meeting ≥ 1 of the following criteria:

  * Clinical stage ≥ T3
  * Gleason score ≥ 8
  * PSA ≥ 20 ng/mL
* Previously untreated disease
* Non-metastatic disease as assessed by bone scan and CT scan of the thorax and abdomen
* Negative pelvic lymph nodes as proven by pathological analysis

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* WBC ≥ 3.5 x 10^9/L
* ANC ≥ 1.5 x 10^9/L
* Platelets normal
* Hemoglobin > 10 g/dL
* Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Albumin ≥ 3 g/dL
* Serum transaminases activity ≤ 2.5 x ULN
* Alkaline phosphatase ≤ 2.5 x ULN
* Serum creatinine ≤ 1.5 x ULN
* Covered by national health insurance
* No history of previous malignant disease, except for adequately treated basal cell carcinoma of the skin
* No ≥ grade 3 hypercholesterolemia/hypertriglyceridemia or ≥ grade 2 hypercholesterolemia/hypertriglyceridemia with history of coronary artery disease (despite lipid-lowering treatment, if given)
* No uncontrolled infection
* No dysphagia or intestinal malabsorption
* No other concurrent severe and/or uncontrolled medical disease that could compromise participation in the study (i.e., uncontrolled diabetes mellitus, uncontrolled cardiac disease [unstable angina], uncontrolled hypertension, congestive cardiac failure, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within the past six months, chronic liver or renal disease, and active upper gastrointestinal tract ulceration)
* No history of noncompliance to medical regimens
* No known hypersensitivity to everolimus, sirolimus (rapamycin), or temsirolimus
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study treatment and follow-up schedule

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 30 days since prior investigational drugs
* More than 10 days since prior and no concurrent treatment with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Acute and late toxicities | 1 year

SECONDARY OUTCOMES:
Biochemical-free survival | 1 year
Metastasis-free survival | 1 year
Overall survival | 1 year
Pre-treatment molecular characteristics of the tumor and its correlation with outcomes | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David Azria, MD, PhD, Principal Investigator — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France